CLINICAL TRIAL: NCT04680689
Title: Assessment of Lesion-Associated Myocardial Ischemia Based on Fusion Coronary CT Imaging- the FUSE-HEART Study: Protocol for a Non-randomised Clinical Trial
Brief Title: Assessment of Lesion-Associated Myocardial Ischemia Based on Fusion Coronary CT Imaging
Acronym: FUSE-HEART
Status: Completed | Type: Observational
Sponsor: Cardio Med Medical Center (Industry)
Collaborators: George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures (Other); Tîrgu Mureș Emergency Clinical County Hospital, Romania (Other)
Responsible Party: Sponsor
Other Study IDs: CM0520-FUSEH
Record Dates: First submitted 2020-12-14; First posted 2020-12-23 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-02

CONDITIONS: Myocardial Ischemia; Myocardial Viability; Coronary Stenosis; Vulnerable Coronary Plaques
Keywords: Fusion imaging; CCTA; Myocardial viability; Vulnerable coronary plaques
MeSH Terms: conditions — Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venous blood samples for complete blood count, biochemistry, inflammatory biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fuse-Heart -SG 01: Study subjects with anatomically significant coronary lesions (at least 50% luminal narrowing) on native coronary arteries.
  Interventions: Diagnostic Test: 128 Multislice CT coronary angiography; Diagnostic Test: 2D Cardiac Transthoracic Echocardiography; Diagnostic Test: Laboratory Blood tests
- Fuse-Heart -SG 02: Study subjects surviving an acute myocardial infarction, revascularized or not.
  Interventions: Diagnostic Test: 128 Multislice CT coronary angiography; Diagnostic Test: 2D Cardiac Transthoracic Echocardiography; Diagnostic Test: Laboratory Blood tests

INTERVENTIONS:
Diagnostic Test: 128 Multislice CT coronary angiography — 128 Multislice CT coronary angiography with the evaluation of coronary stenosis, the plaque vulnerability markers ( necrotic core, low attenuation plaque, spotty calcifications, napkin ring sign, positive remodeling), asses polar maps of the myocardium
  Other Names: CCTA
Diagnostic Test: 2D Cardiac Transthoracic Echocardiography — 2D Cardiac Transthoracic Echocardiography with the evaluation of the cardiac cavity dimensions
Diagnostic Test: Laboratory Blood tests — Laboratory tests for evaluations the level of inflammatory biomarkers ( hs-CRP, MMP, IL6 and NT-pro-BNP), complete blood count, biochemestry

SUMMARY:
The aim of the Fused-Heart study is to investigate the impact of a coronary artery stenosis on myocardial function and viability, based on advanced fusion imaging techniques derived from CCTA.

Moreover the study will investigate the correlation between morphology and composition of atheromatous plaques located in a coronary artery and myocardial ischemia in the territory irrigated by the same coronary artery.

DETAILED DESCRIPTION:
The FUSE-HEART study is a prospective, observational, single-center, cohort study that will be conducted in the Laboratory of Advanced Research in Cardiac Multimodal Imaging of Cardio Med Medical Center Targu Mures, Romania.

The study will include 100 subjects with coronary lesions depicted by CCTA examination. The study population will consist in: (1) patients with anatomically significant coronary lesions (at least 50% luminal narrowing) on native coronary arteries, or (2) patients surviving an acute myocardial infarction, revascularized or not. In all patients, presence of vulnerability features in the atheromatous plaques will be studied and the vulnerability score will be calculated for each plaque, consisting in one point added for each of the following vulnerability markers: positive remodeling, napkin-rink sign, presence of low density plaque or spotty calcium within the plaque. In addition, following 3D fusion of the images of the coronary tree with the images reflecting wall motion, the correspondence between plaque morphology and composition on one hand, and wall motion in the corresponding distribution territory of that coronary artery, will be studied based on fused models.

The study will be conducted over a period of 2 years, in which patients will be examined at baseline, with a projected recruitment period of 1 year and will be followed-up 1 year for MACE.

Study objectives:

Primary: to investigate the impact of a coronary artery stenosis on myocardial function and viability, based on advanced fusion imaging techniques derived from CCTA.

Secondary: to investigate the correlation between morphology and composition of atheromatous plaques located in a coronary artery and myocardial ischemia in the territory irrigated by the same coronary artery.

Study timeline:

• Baseline (day 0)-Obtain and document consent from participant on study consent form.

Verify inclusion/exclusion criteria. Obtain demographic information, medical history, medication history, alcohol and tobacco use history. Record results of physical examinations and 12-lead ECG.Collect blood specimens (complete blood count, biochemistry and inflammatory biomarkers).Imaging procedures: CCTA-Image processing - quantification of coronary stenosis, characterization of vulnerability markers, 3D reconstruction, extension and characterization of wall motion. Deliver fused 3D images

• Visit 1 (month 1)-Record results of physical examinations, 12-lead ECG, blood pressure, and medical history. MACE assessment Visit 2 (month 3) -Telephone visit with target questions, all the answers recorded in study forms Visit 3 (month 6) - Record results of physical examinations, 12-lead ECG, blood pressure, and medical history. MACE assessment

Final study visit (month 12)- Record results of physical examinations, medical history,12-lead ECG, blood pressure, transthoracic 2-D echocardiography. End-point and MACE evaluation.

Study procedures:

* Medical history, clinical examination, laboratory tests (complete blood count, biochemistry, inflammatory biomarkers: hs-CRP, MMP, IL6 and NT-pro-BNP);
* 12-lead ECG
* 2D transthoracic echocardiography
* CCTA
* Computerized postprocessing and fused images

Data collection:

All the information will be collected in a dedicated database including medical history, medication, imaging features provided by cardiac ultrasound, CCTA and fused images resulting from imaging post-processing.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CCTA examination, with at least one coronary artery lesion producing a luminal narrowing >50%
* Ability to provide informed consent;
* Patients aged at least 18 years;

Exclusion Criteria:

* Unwillingness or incapacity to provide informed consent;
* Allergy to contrast media;
* Absolute or relative contraindications to CCTA imaging;
* Irregular or rapid heart rhythm
* Pregnancy or lactation;
* Women with childbearing potential in absence of any contraceptive treatment;
* Renal insufficiency (creatinine greater than 1.5 mg/dL) or renal failure requiring dialysis;
* Active malignancy or malignancy within the last 5 year prior to enrollment;
* Conditions associated with an estimated life expectancy of under 2 years;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 100 subjects with coronary lesions depicted by CCTA examination. The study population will consist in: (1) patients with anatomically significant coronary lesions (at least 50% luminal narrowing) on native coronary arteries, or (2) patients surviving an acute myocardial infarction, revascularized or not.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
MACE rate-Major Adverse Cardiovascular Events | 12 months
  The primary outcome of the study is represented by the rate of MACE events related to myocardial ischemia at 1-year post assessment, in correlation with the degree of coronary artery stenosis and myocardial ischemia or viability.

SECONDARY OUTCOMES:
Re-hospitalisation rate, | 12 months
  Secondary outcome refers to rate of re-hospitalization, in correlation with the morphology and composition of atheromatous plaques located in a coronary artery and myocardial ischemia in the territory irrigated by the same coronary artery
Rate of survival | 12 months
  This outcome refers to rate of survival in correlation with the morphology and composition of atheromatous plaques located in a coronary artery and myocardial ischemia in the territory irrigated by the same coronary artery

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Gorea Stanescu, MD, Principal Investigator — Cardio Med
Locations (1):
- Cardio Med Medical Center, Târgu Mureş, Mureș County, Romania

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available for interested parties
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The IPD sharing time is starting 6 months aflter publication